CLINICAL TRIAL: NCT02038374
Title: Clinico-biological Correlation of Severe Asthma in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2013-A00401-44; 2013-06 (Other: AP HM)
Record Dates: First submitted 2013-09-12; First posted 2014-01-16 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- severe asthma atopic (Experimental)
  Interventions: Procedure: biopsies
- asthma non atopic (Experimental)
  Interventions: Procedure: biopsies

INTERVENTIONS:
Procedure: biopsies

SUMMARY:
Asthma is the most common chronic respiratory disorder in children. Despite significant advances in understanding of asthma, available therapies fail to alter the natural history and progression of the disease. Airway epithelial cells are continuously exposed to and injured by environmental irritants, such as viruses and pollutants, and as such are ideally situated to orchestrate airway function in response to these stimuli.

Severe or difficult-to-treat asthma in children is a complicated disorder characterized by ongoing symptoms and persistent airway inflammation and oxidant stress despite corticosteroid treatment. Although severe asthma is likely a heterogeneous disorder, affected children similar clinical features, including gas trapping, bronchial hyperresponsiveness, and aeroallergen sensitization. However, the molecular and cellular pattern of inflammation in children with severe asthma are not uniform : some investigators have found increased eosinophils and TH2 derived cytokines, others have noted noneosinophilic patterns with neutrophil activation.

Given the heterogeneity of the inflammatory response in children with severe asthma, additional methods to distinguish severe asthma are needed.

ELIGIBILITY:
Inclusion Criteria:

* Children 0-18 years
* patients followed regularly for at least one year.
* The diagnosis of asthma is increased according to the criteria of the Global Initiative for Asthma (GINA): children with a history of recurrent episodes of bronchial obstruction.
* children with severe asthma defined by the American Thoracic Society (ATS): Severe asthma is defined by the presence of a major criterion: the need for high doses of inhaled corticosteroids (budesonide dose equivalent 400 micro g) and least two of the five minor criteria:
* The daily use of beta 2 long-acting or short-term daily action (<4 years) or anti-leukotrienes associated with inhaled corticosteroids Daily or almost daily use of beta-2 short-acting Permanent-bronchial obstruction (FEV <80% predicted FEV)
* At least one emergency department visit for asthma exacerbations in France
* At least 3 courses of oral corticosteroids per year

Exclusion Criteria:

* parents' refusal to participate in the study
* refusal children to participate pathology underlying cardiac, neuromuscular, immunodeficiency

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-09 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
analysis of bronchial biopsies | 12 months
  Number of ciliated cells(units) versus cells(units) with mucus found by fields of interface of the culture

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France